CLINICAL TRIAL: NCT03399955
Title: An Open Label, Randomized, Parallel Arm Clinical Trial of Two Regimens to Assess the Safety and Efficacy for Treatment of Post Kala-azar Dermal Leishmaniasis (PKDL) Patients in Sudan
Brief Title: Short Course Regimens for Treatment of PKDL (Sudan)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-MILT COMB-02-PKDL
Record Dates: First submitted 2017-12-07; First posted 2018-01-17 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: PKDL - Post-Kala-Azar Dermal Leishmanioid
MeSH Terms: interventions — Paromomycin; liposomal amphotericin B; miltefosine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Paromomycin + Miltefosine (Experimental): Paromomycin 20 mg/kg/d IM for 14 days combined with Miltefosine allometric BID PO dosing for 42 days
  Interventions: Drug: Paromomycin; Drug: Miltefosine
- Arm 2: Ambisome + Miltefosine (Experimental): AmBisome® 5mg/kg/d IV infusion at D1, D3, D5 and D7 (20 mg/kg total dose) combined with Miltefosine allometric BID PO dosing for 28 days
  Interventions: Drug: Ambisome; Drug: Miltefosine

INTERVENTIONS:
Drug: Paromomycin — Paromomycin (20 mg/kg/d) IM for 14 days
  Arms: Arm 1: Paromomycin + Miltefosine
Drug: Ambisome — AmBisome® (20 mg/kg total dose) IV over 7 days
  Other Names: Liposomal Amphotericin B
  Arms: Arm 2: Ambisome + Miltefosine
Drug: Miltefosine — Miltefosine oral (allometric dosing) for 42 days (arm 1) or 28 days (arm 2)
  Other Names: Impavido

SUMMARY:
This is an open label, randomized non comparative phase II clinical trial conducted on parallel groups, to assess the safety and efficacy of the combination of Paromomycin (20 mg/kg/d) IM for 14 days and Miltefosine (allometric dosing) oral for 42 days, and a combination of AmBisome® (20 mg/kg total dose) IV over 7 days and Miltefosine oral for 28 days (allometric dosing) for the treatment of PKDL patients in Sudan.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PKDL case by clinical presentation and demonstration of parasites by microscopy in a skin smear or by PCR, with documented stable or progressive disease for at least 6 months or grade 3 PKDL
* Male or Female patients aged 6 to 60 years
* Written voluntarily informed consent is obtained from the patient, or his guardian if the patient is < 18 years old. In the case of minors aged >12 to <18, assent from the children is also needed in addition to the guardian's consent.

Exclusion Criteria:

* Patients who had prior treatment of PKDL within the last 1 year
* Pregnant and lactating women and women of childbearing age (12 to 55 years) who do not accept to have a pregnancy test and who do not agree to use contraception during treatment period and for 5 months after the end of treatment.
* Patients with signs and symptoms of severe diseases: defined as suffering from a concomitant severe infection such as TB or any other serious known underlying disease (cardiac, renal, hepatic),
* Severe malnutrition defined by BMI for age WHO reference curves for gender, Z score < -3 for subjects 6 to < 19 years; BMI < 16 for subjects > 19 years old
* Patients with haemoglobin < 5g/dL
* Patients with known skin disease
* Patients with abnormal liver function (ALT and AST) tests of more than three times the normal range.
* Patients with total bilirubin levels >1.5 times the upper normal range
* Patients with serum creatinine above the upper limit of normal range
* Patients with serum potassium < 3.5 mmol/L
* Patients with pre-existing clinical hearing loss based on audiometry at baseline
* Patients with a positive HIV test as applicable
* Patients / guardian not willing to participate
* Patients with history of allergy or hypersensitivity to the relevant study drug
* Patients on immunomodulators therapy

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-05-09 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Definitive Cure | 12 months follow-up assessment
  definitive cure at 12 months after treatment onset, defined as clinical cure (100% lesions resolution) and no additional PKDL treatment between end of therapy and 12 months follow-up assessment.
Incidence of treatment-emergent adverse events | from start of treatment to 12 month follow-up
  Frequency of SAE from start of treatment to 12 months follow-up Frequency and severity of all adverse events Frequency and severity of adverse events that lead to treatment discontinuation

SECONDARY OUTCOMES:
Pharmacokinetics of Miltefosine | Miltefosine concentration in the skin will be measured at day 14 and day 42 for MF+PM arm and at day 7 and day 28 for Ambisome+MF arm. Miltefosine concentration in the blood will be measured at day 1, day 7, day 14, day 28, day 42 and 3 month
  To assess the maximal accumulation (Cmax) of Miltefosine in the skin at the end of treatment and correlate it with achieved plasma concentrations.
Pharmacokinetics of Amphotericin B (MF + Ambisome arm only) | Amphotericin B concentration will be measured in the skin at day 7 and day 28. Amphotericin B concentration in the blood will be measured at day 1 and day 7.
  To assess the maximal accumulation (Cmax) of Amphotericin B in the skin at the end of treatment and correlate it with achieved plasma concentrations.
Pharmacokinetics of Paromomycin (MF + Paromomycin arm only) | Paromomycin concentration will be measured in the skin at day 14 and day 42. Paromomycin concentration in the blood will be measured at day 1 and day 14.
  To assess the maximal accumulation (Cmax) of Paromomycin in the skin at the end of treatment and correlate it with achieved plasma concentrations.
Immune Response | At screening, at day 42 (end of treatment) and at 6 month follow-up
  To assess the change in immune response during and after end of treatment by measuring cytokines profiles level in the peripheral blood.
Parasite quantification in blood and skin | At screening, day 42 (end of treatment), 3 month follow-up, 6 month follow-up and 12 month follow-up.
  Parasites will be quantified in blood and skin, by microscopy and qPCR, to assess the clearance before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Elhassan Centre for tropical Medicine, Doka, Al Qaḑārif, Sudan

REFERENCES:
- [Derived] Torres A, Younis BM, Alamin M, Tesema S, Bernardo L, Solana JC, Moreno J, Mustafa AA, Alves F, Musa AM, Carrillo E. Differences in the Cellular Immune Response during and after Treatment of Sudanese Patients with Post-kala-azar Dermal Leishmaniasis, and Possible Implications for Outcome. J Epidemiol Glob Health. 2024 Sep;14(3):1167-1179. doi: 10.1007/s44197-024-00270-0. Epub 2024 Jul 15. PMID 39007942
- [Derived] Younis BM, Mudawi Musa A, Monnerat S, Abdelrahim Saeed M, Awad Gasim Khalil E, Elbashir Ahmed A, Ahmed Ali M, Noureldin A, Muthoni Ouattara G, Nyakaya GM, Teshome S, Omollo T, Ochieng M, Egondi T, Mmbone M, Chu WY, Dorlo TPC, Zijlstra EE, Wasunna M, Alvar J, Alves F. Safety and efficacy of paromomycin/miltefosine/liposomal amphotericin B combinations for the treatment of post-kala-azar dermal leishmaniasis in Sudan: A phase II, open label, randomized, parallel arm study. PLoS Negl Trop Dis. 2023 Nov 21;17(11):e0011780. doi: 10.1371/journal.pntd.0011780. eCollection 2023 Nov. PMID 37988402